CLINICAL TRIAL: NCT04410601
Title: Pre-and Post-operative Risk Factors Affecting the Incidence and Severity of Dysphagia Following Total Thyroidectomy: An International Multi-centric Prospective Randomized Controlled Clinical Trial (RCT)
Brief Title: Post-thyroidectomy Dysphagia: An International Multicentric CONSORT - Compatible RCT
Acronym: Dysphagia-TT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ethem Unal, M.D., PhD, Associate Prof of Surgery & Surgic, Associated Professor of General Surgery and Surgical Oncology, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01/173; 12.05.2020/173 (Registry Identifier: SBU-UmraniyeERH-Ethics Committee-approved RCT)
Record Dates: First submitted 2020-05-15; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Dysphagia, Esophageal; Dysphagia, Oral Phase; Dysphagia Comes and Goes; Thyroiditis; Thyroid Cancer; Thyroid Neoplasms; Thyroid Goiter; Thyroid Nodule (Benign)
Keywords: Thyroidectomy; Total thyroidectomy; Post-thyroidectomy; Post-thyroidectomy dysphagia; International; Multi-centric
MeSH Terms: conditions — Deglutition Disorders; Thyroiditis; Thyroid Neoplasms; Goiter; Thyroid Nodule

STUDY DESIGN:
Intervention Model Description: Dysphagia among patients who have undergone total hyroidectomy for benign/malign thyroid disease. The preoperative factors (demographics; co-morbidities such as diabetes, multiple sclerosis, Parkinson's; body mass index; routine ear-nose-throat-ENT consultation), operative factors (over-manipulation, injury to larynx/neural plexus, easy/hard tracheal intubation, closure of strap muscles/stay open) and postoperative evaluation 1-No dysphagia, 2-Dysphagia with at least one other complication (nerve injury, hypocalcemia), 3-Dysphagia without any other surgical complications; ENT&neurology consultations, survey.
Masking Description: THE STUDY IS OPEN TO ALL SURGICAL CLINICS OVER THE WORLD EAGER TO JOIN; EXCEL WITH FORMS TO BE FILLED ARE AVAILABLE, please contact the principle/co-investigators by phone/e-mail.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No dysphagia (after total thyroidectomy-TT) (Active Comparator): Patients s/p post-thyroidectomy without complication
  *will NOT be enrolled to standard dysphagia-rehabilitation treatment
  Interventions: Procedure: Total thyroidectomy
- Dysphagia (with at least one more complication of TT) (Experimental): Patients s/p post-thyroidectomy with both dysphagia and other documented TT complication such as vocal cord paralysis/hypocalcemia/surgical site infection etc.
  *will be enrolled to standard dysphagia-rehabilitation treatment for 6-week.
  Interventions: Procedure: Total thyroidectomy
- Dysphagia (the only complication after TT) (Experimental): Patients s/p post-thyroidectomy dysphagia only.
  *will be enrolled to standard dysphagia-rehabilitation treatment for 6-week.
  Interventions: Procedure: Total thyroidectomy

INTERVENTIONS:
Procedure: Total thyroidectomy — DRT-diet modification, compensation strategies, oral motor exercises such as laryngeal elevation, masseters / tongue hold / exercise, bolus transition exercise; chin-down/up, head rotation, and other maneuvers with tactile stimulation.
  Other Names: Dysphagia rehabilitation treatment (DRT) programme

SUMMARY:
The most common and feared complications of total thyroidectomy are vocal cord paralyses and hypocalcemia. However, post-thyroidectomy dysphagia is not uncommon and has important consequences on the quality of life (QoL). It should be taken seriously by all clinicians.

DETAILED DESCRIPTION:
Dysphagia is a possible complication that can be observed in patients undergoing thyroidectomy, and can be related to superior and inferior laryngeal nerves dysfunction, but it usually appears after an uncomplicated surgical procedure. Aerodigestive symptoms, such as discomfort, tightness, lump, foreign body, difficulty or pain during swallowin, can also present before operation. If it appears or aggrevates after surgery, laryngeal nerve damage (superior laryngeal nerve - SLN, or inferior laryngeal nerve - recurrent, RLN), tracheo-malacia and postoperative fibrotic changes should be interrogated. However, in most of the cases, an anatomic and/or physiologic defect in the oro-pharngeal region is not easy to be detected. Therefore, a subjective feeling of dysphagia is more common.

Dysphagia has important consequences on the QoL in postoperative period, and should be addressed by the primary surgeon/clinician, regardless of whether it is objective or subjective.

The goal of the present study is to better understand the incidence of postoperative dysphagia symptoms among patients who have undergone total thyroidectomy for benign or malign thyroid disease. Besides, all possible risk factors (pre-intra-post-operative) are also going to be evaluated in detail, and the efficacy of a 6-week dysphagia-rehabilitation programme will also be employed and results will be shared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with benign or malignant thyroid disorder (multinodular goitre, toxic goitre, thyroid carcinoma)
* Patients with total thyroidectomy (TT) indication
* Patients over 17 year-old

Exclusion Criteria:

* Patients without thyroid disease
* Patients with thyroid disorder, but prepared for surgery other than TT
* Healthy volunteers
* Patients below 17 y/o

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Dysphagia-Subjective Survey Form | 12 months
  Subjective survey form to be filled- a self-evaluation questionnaire-to evaluate 'Change from baseline postoperative (po) day 1-3 to week 2, po week 6, po week 16, po week 24, po week 36 and po week 48 (last). A new form will be filled in for each outpatient clinic control.
  assessing common dysphagia symptoms- includes 6 items scored within a range of 0 (without swallowing alterations) to 24 (maximum swallowing dysfunction).
Evaluation of Dysphagia-Objective Functional Outcome Swallowing Score (FOSS) | 12 months
  Objective survey form to be filled- a clinician-oriented questionnaire assessing the swallowing function objectively, from stage I (normal function) to stage V (no oral intake). To evaluate change in dysphagia from baseline po day 1-3 to .po week 2, po week 6, po week 16, po week 24, po week 36 and po week 48 (last). A new form will be filled in for each outpatient clinic control.
Evaluation of Dysphagia- ENT Consultation | 12 months
  Flexible fiberoptic laryngoscopy (any anatomic explanation for dysphagia? YES or NO? To evaluate change in dysphagia from baseline at postoperative (po) week 6 to po week 24, po week 48 (last).
Evaluation of Dysphagia- Neurology Consultation | 12 months
  EMG-electromyography test (any anatomic and/or physiologic dysfunction? YES or NO? To evaluate change in dysphagia from baseline at postoperative (po) week 6 to po week 24, po week 48 (last).
Evaluation of Dysphagia- Esophago-gastro-duodenoscopy (EGD) | 6 weeks
  Any anatomic defect? EGD will be performed once at Postoperative (po) week 6.

SECONDARY OUTCOMES:
Evaluation of Standard Dysphagia Rehabilitation | 12 weeks
  6-week treatment, starting from po week 6, for all patients with dysphagia- ending at po week 12. Any improvement after 6-week treatment? evaluate at po week 12 and please answer: Any improvent in dysphagia symptom? -YES or NO?

CONTACTS AND LOCATIONS:
Overall Officials: Sema YUKSEKDAG, MD, Principal Investigator — Instructor in General Surgery; Ethem UNAL, MD, PhD, ECFMG, IFSO & Board CSS, Study Chair — Assoc. Professor of General Surgery and Surgical Oncology
Locations (1):
- Umraniye Education and Research Hospital, Health Sciences University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Excel documents including data (patient ID and protocol # will be shaded) available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months from the beginning (01.06.2020)
Access Criteria: All surgical clinics/Investigators are WELCOME / INVITED to join this CONSORT-compatible RCT
URL: http://www.consort-statement.org/

REFERENCES:
- [Background] Rihn JA, Kane J, Albert TJ, Vaccaro AR, Hilibrand AS. What is the incidence and severity of dysphagia after anterior cervical surgery? Clin Orthop Relat Res. 2011 Mar;469(3):658-65. doi: 10.1007/s11999-010-1731-8. PMID 21140251
- [Background] Hashemian M, Khorasani B, Tarameshlu M, Haghani H, Ghelichi L, Nakhostin Ansari N. Effects of Dysphagia Therapy on Swallowing Dysfunction after Total Thyroidectomy. Iran J Otorhinolaryngol. 2019 Nov;31(107):329-334. doi: 10.22038/ijorl.2019.36233.2193. PMID 31857976
- [Background] Exarchos ST, Lachanas VA, Tsiouvaka S, Tsea M, Hajiioannou JK, Skoulakis CE, Bizakis JG. The impact of perioperative dexamethasone on swallowing impairment score after thyroidectomy: a retrospective study of 118 total thyroidectomies. Clin Otolaryngol. 2016 Oct;41(5):615-8. doi: 10.1111/coa.12547. Epub 2016 Feb 8. No abstract available. PMID 26434490
- [Background] Shimizu M, Kobayashi T, Jimbo S, Senoo I, Ito H. Clinical evaluation of surgery for osteophyte-associated dysphagia using the functional outcome swallowing scale. PLoS One. 2018 Aug 1;13(8):e0201559. doi: 10.1371/journal.pone.0201559. eCollection 2018. PMID 30067834
- [Result] Scerrino G, Tudisca C, Bonventre S, Raspanti C, Picone D, Porrello C, Paladino NC, Vernuccio F, Cupido F, Cocorullo G, Lo Re G, Gulotta G. Swallowing disorders after thyroidectomy: What we know and where we are. A systematic review. Int J Surg. 2017 May;41 Suppl 1:S94-S102. doi: 10.1016/j.ijsu.2017.03.078. PMID 28506421
- See also: Ethem Unal, MD, PhD, ECFMG, IFSO, BCSS, Assoc. Professor of General Surgery & Surgical Oncology, H-index:18 / i10-index:33 — https://scholar.google.com.tr/citations?user=6bFlCZwAAAAJ&hl=tr